CLINICAL TRIAL: NCT01792921
Title: COG FUN Intervention for ADHD
Brief Title: Effectiveness of a Cognitive-functional (Cog-Fun) Intervention for Children With ADHD
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, BERGER ITAI, Director, Neurocognitive Center HMO, Hadassah Medical Organization
Other Study IDs: HMO-0576-12
Record Dates: First submitted 2013-01-27; First posted 2013-02-15 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: ADHD
Keywords: Age 7-10 years old; regular education system; no moderate or severe neurological and/or psychiatric disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- control waitlist
  Interventions: Behavioral: COG - FUN

INTERVENTIONS:
Behavioral: COG - FUN

SUMMARY:
Scientific Rationale: Many children with ADHD have serious difficulties in participation in daily occupations in their ecological settings. These difficulties have a pervasive negative impact on their everyday functioning and quality of life (QoL). Although pharmacological treatment has been proven effective in treating ADHD symptoms in many children, as have psychosocial interventions such as parent training, there is little evidence for integrative approaches that address the cognitive, volitional and social-environmental barriers to participation with this population. Although preliminary positive effects of a cognitive-function (Cog-Fun) treatment in occupational therapy on this population have been demonstrated, additional evidence is needed to confirm these initial findings. Methods: Initial results of our pilot study (N=17 children with ADHD) demonstrated significant moderate to large effects of Cog-Fun treatment, which targeted participation and executive functions in daily life. Significant effects were also found for a measure of self-efficacy and neuropsychological measures of attention, planning and organization. Parent ratings showed significant reduction of ADHD symptoms and improved QoL. The purpose of the current study is to replicate the pilot study findings in a randomized controlled trial. The study will be a randomized controlled trial with a crossover design, including 2 groups of children with ADHD attending elementary school and their parents. The research group (Group A, n=50) will receive three months of the Cog-Fun treatment, designed for a parent/child dyad and the control group (Group B, n=50) will be wait-listed and receive treatment after three months. Outcomes will include measures of participation, executive functions in daily life, child and parental self-efficacy, ADHD symptoms and QoL. The investigators expect to find a significant main effect of time (pre-post intervention), group (research vs. control) and a significant interaction effect (group x time) on executive and occupational outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ADHD
* 7-10 years old
* regular education system
* no moderate or severe neurological and/or psychiatric disorders

Exclusion Criteria:

* moderate or severe neurological and/or psychiatric disorders

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children age 7-10 years diagnosed with ADHD
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in ADHD parameters | Three assessment points - at recruitment, after 3 months and after 6 months.
  Using Brief Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Hahn-Markowitz J, Manor I, Maeir A. Effectiveness of cognitive-functional (Cog-Fun) intervention with children with attention deficit hyperactivity disorder: a pilot study. Am J Occup Ther. 2011 Jul-Aug;65(4):384-92. doi: 10.5014/ajot.2011.000901. PMID 21834453